CLINICAL TRIAL: NCT02229253
Title: Real-life Data of Cardiovascular Events Occuring During Degarelix Therapy for Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000171
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Advanced Hormone Sensitive Prostate Cancer
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Degarelix: Treatment according to standard clinical practice.
  Interventions: Drug: degarelix

INTERVENTIONS:
Drug: degarelix
  Other Names: Firmagon®

SUMMARY:
Patients with prostate cancer and a history of cardiovascular disease treated with degarelix for their prostate cancer, will be followed for a period of one year. In this real-life, non-interventional trial, any cardiovascular events occurring during degarelix therapy will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer and a history of cardiovascular disease, prescribed degarelix for the treatment of their prostate cancer

Exclusion Criteria:

* Patients who have received a form of androgen deprivation therapy for their prostate cancer, during the 12 months preceding this study are excluded
* Planned intermittent or short-term (< 12 months) degarelix treatment
* Planned addition of, or switch to another form of androgen deprivation therapy during the study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected from prostate cancer patients in a hospital setting, meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular event rate in hormone naïve prostate cancer patients with cardiovascular comorbidity at baseline, treated with degarelix in daily practice | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Groene Hart Ziekenhuis (there may be other sites in this country), Gouda, Netherlands